CLINICAL TRIAL: NCT05443451
Title: 3D-Ultrasound-Guided Transperineal Microwave Needle Ablation for Men With Symptomatic Benign Prostatic Hyperplasia
Brief Title: BETTY: BEnign Prostatic Hyperplasia Transperineal Targeted Microwave therapY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Koelis (Industry)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2022.249
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transperineal Microwave needle ablation for symptomatic BPH (Experimental)
  Interventions: Device: 3D-Ultrasound-Guided Transperineal Microwave needle ablation of BPH

INTERVENTIONS:
Device: 3D-Ultrasound-Guided Transperineal Microwave needle ablation of BPH — The procedure will consist of a focal, transperineal, targeted microwave ablation of prostate adenoma. Surgical planning using 3D transrectal ultrasound and real-time monitoring of the ablation would preserve key anatomical landmarks such as the bladder neck, prostatic urethra and verumontanum. The Organ-Based Tracking (OBT®) patented technology would provide a 3D prostate model to facilitate real-time navigation-guided ablation and accurate mapping of treatment zone. The procedure will be conducted under general anaesthesia, spinal anaesthesia, or monitored anaesthetic care / sedation. An average number of one to three microwave ablations per lobe is expected, depending on the size and shape of each prostate. The microwave ablation parameters will be chosen intraoperatively. A urinary catheter may be necessary immediately after the procedure. Patients are planned to be discharged on the same day or the day after when they are fit for discharge.

SUMMARY:
This is a pilot study on applying 3D-Ultrasound-Guided Transperineal Microwave needle ablation for men with symptomatic benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
This is a prospective, single centre, open-label and non-comparative trial planned on 12 patients. Patients who fit inclusion criteria would be recruited and offered microwave ablation to the enlarged prostate. The patients will be closely followed up to 6 months after treatment with serial assessment on safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years.
* Benign prostatic hyperplasia with prostate size 30-80 cc
* IPSS ≥ 14
* PSA ≤ 4 ng/mL or PSA >4 ng/mL with no evidence of suspicious lesion on mpMRI
* Maximum urine flow rate (Qmax) ≤ 15 mL/s.
* Post-Void Residual ≤ 150 mL.
* Patient suitable for IV sedation and/or spinal anaesthesia and/or general anaesthesia and focal microwave ablation.
* Informed written consent

Exclusion Criteria:

* Significant intravesical median lobe hyperplasia.
* Suspicious lesion on mpMRI prostate
* History of prostate, bladder or urethral surgery.
* History of prostate cancer
* Presence of stones, bladder diverticulum and/or bladder tumor
* History of long-term indwelling catheter.
* Urethral stricture
* Known coagulopathy or on anticoagulant
* Presence of a pacemaker.
* Active infection
* Dysuria due to bladder dysfunction.
* Serious medical illness, including any of the following: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction, cerebrovascular event within 6 months prior to the screening visit.
* Neurological disorders that would impact bladder function (e.g., multiple sclerosis, Parkinson's disease, spinal cord injury).
* Contraindications for mpMRI exam or MR contrast
* Acute and/or chronic renal failure (GFR <50 ml/min and serum creatinine > 1.5 mg/d).
* Patient currently participating in another interventional clinical trial.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with prostate
Enrollment: 12 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) and serious adverse events (SAE) related to the treatment | At 1 month
  The severity of AE is grade by Clavien-Dindo classification.

SECONDARY OUTCOMES:
Prostate volume change | Baseline, 3 months, 6 months
  Prostate volume change after treatment
Urinary symptoms measured by International Prostate Symptom Score (IPSS) score | Baseline, 1 month, 3 months, 6 months
  Change in total scores in International Prostate Symptom Score (ranges from 0 to 35) questionnaires. The higher score, the more worse symptom.
Erectile function measured by International Index of Erectile Function 5-item version (IIEF-5) score | Baseline, 1 month, 3 months, 6 months
  Change in International Index of Erectile Function 5 questionnaire score (ranges from 0 to 25). The higher score, the more worse symptom.
Ejaculatory function measured by MSHQ-EjD-SF (function and bother) score | Baseline, 1 month, 3 months, 6 months
  Change in MSHQ-EjD-SF questionnaire score (Range from 1-15 for function and and 0-5 for bother). The higher score, the more worse symptom.
Change in urodynamic in uroflowmetry | Baseline, 1 month, 3 months, 6 months
  Change in urodynamic function assessed by uroflowmetry, parameters include voided volume, maximum flow rate and post-void residual.
PSA change | Baseline, 3 months, 6 months
  PSA change after treatment
Average patient post-operative pain level | Baseline, 2 and 4 hours after the procedure and at 1-week
  Assessed by a pain numeric rating scale, Score 0-10, the higher score the worsen pain
Patient quality of life | Baseline, 1-week, 1-month, 3-month, and 6-month,
  Assessed with the EQ-5D-5L questionnaire, the higher the score the better in quality of life
Patient satisfaction | Baseline, 1-week, 1-month, 3-month, and 6-month,
  Assessed with the PGI-I questionnaire,the lower score the more satisfaction
Ease of the procedure measured with a score chosen by the operator | Post procedure immediately
  1: easy, 2: moderate, 3: difficult
Ablation treatment time | Intra-operation
  Duration of the ablation procedure
Length of hospital stay | The total number of days of hospitalization for this surgical procedure up to day 30 after the procedure]
  Total number of days of hospitalization for the surgical procedure
Operation time | Intra-operation
  Duration of patients stay in Operation Room

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fung CHIU, FRCS, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Zhang X, Li H, Wu F, Wang H, Zhao M, Hu H, Xu K. Prevalence of lower urinary tract symptoms suggestive of benign prostatic hyperplasia (LUTS/BPH) in China: results from the China Health and Retirement Longitudinal Study. BMJ Open. 2019 Jun 19;9(6):e022792. doi: 10.1136/bmjopen-2018-022792. PMID 31221864
- [Background] Roehrborn CG, Siami P, Barkin J, Damiao R, Major-Walker K, Nandy I, Morrill BB, Gagnier RP, Montorsi F; CombAT Study Group. The effects of combination therapy with dutasteride and tamsulosin on clinical outcomes in men with symptomatic benign prostatic hyperplasia: 4-year results from the CombAT study. Eur Urol. 2010 Jan;57(1):123-31. doi: 10.1016/j.eururo.2009.09.035. Epub 2009 Sep 19. PMID 19825505
- [Background] Ng CF, Yee CH, Chan CK, Wong HM, Chiu PK, Tsu JH, Teoh JY, Ho KL. Bipolar transurethral vapourisation versus monopolar transurethral resection of prostate: a randomised controlled trial. Hong Kong Med J. 2017 Jun;23 Suppl 2(3):32-34. No abstract available. PMID 29938669
- [Background] Yee CH, Wong JH, Chiu PK, Chan CK, Lee WM, Tsu JH, Teoh JY, Ng CF. Short-stay transurethral prostate surgery: A randomized controlled trial comparing transurethral resection in saline bipolar transurethral vaporization of the prostate with monopolar transurethral resection. Asian J Endosc Surg. 2015 Aug;8(3):316-22. doi: 10.1111/ases.12197. Epub 2015 Jun 3. PMID 26042336
- [Background] Madersbacher S, Lackner J, Brossner C, Rohlich M, Stancik I, Willinger M, Schatzl G; Prostate Study Group of the Austrian Society of Urology. Reoperation, myocardial infarction and mortality after transurethral and open prostatectomy: a nation-wide, long-term analysis of 23,123 cases. Eur Urol. 2005 Apr;47(4):499-504. doi: 10.1016/j.eururo.2004.12.010. Epub 2005 Jan 23. PMID 15774249
- [Background] Raizenne BL, Zheng X, Mao J, Zorn KC, Cho A, Elterman D, Bhojani N, Sedrakyan A, Chughtai B. Real-world data comparing minimally invasive surgeries for benign prostatic hyperplasia. World J Urol. 2022 May;40(5):1185-1193. doi: 10.1007/s00345-021-03926-9. Epub 2022 Feb 2. PMID 35107632
- [Background] Chughtai B, Elterman D, Shore N, Gittleman M, Motola J, Pike S, Hermann C, Terrens W, Kohan A, Gonzalez RR, Katz A, Schiff J, Goldfischer E, Grunberger I, Tu LM, Alshak MN, Kaminetzky J. The iTind Temporarily Implanted Nitinol Device for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia: A Multicenter, Randomized, Controlled Trial. Urology. 2021 Jul;153:270-276. doi: 10.1016/j.urology.2020.12.022. Epub 2020 Dec 26. PMID 33373708
- [Background] McVary KT, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Pliskin M, Beahrs JR, Prall D, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Tadros NN, Gange SN, Roehrborn CG. Final 5-Year Outcomes of the Multicenter Randomized Sham-Controlled Trial of a Water Vapor Thermal Therapy for Treatment of Moderate to Severe Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2021 Sep;206(3):715-724. doi: 10.1097/JU.0000000000001778. Epub 2021 Apr 19. PMID 33872051
- [Background] Chiu PK, Lo KL, Teoh JY, Ma SF, Leung CH, Wong HF, Li KM, Sae-Lo K, Kwok SW, Li SY, Yee CH, Hou SM, Ng CF. Sectoral cancer detection and tolerability of freehand transperineal prostate biopsy under local anaesthesia. Prostate Cancer Prostatic Dis. 2021 Jun;24(2):431-438. doi: 10.1038/s41391-020-00293-1. Epub 2020 Sep 30. PMID 32999465
- [Background] Barry Delongchamps N, Schull A, Anract J, Abecassis JP, Zerbib M, Sibony M, Jilet L, Abdoul H, Goffin V, Peyromaure M. Feasibility and safety of targeted focal microwave ablation of the index tumor in patients with low to intermediate risk prostate cancer: Results of the FOSTINE trial. PLoS One. 2021 Jul 14;16(7):e0252040. doi: 10.1371/journal.pone.0252040. eCollection 2021. PMID 34260598
- [Background] Lo KL, Chui KL, Leung CH, Ma SF, Lim K, Ng T, Wong J, Li JKM, Mak SK, Ng CF. Outcomes of transperineal and transrectal ultrasound-guided prostate biopsy. Hong Kong Med J. 2019 Jun;25(3):209-215. doi: 10.12809/hkmj187599. Epub 2019 May 29. PMID 31178436
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542